CLINICAL TRIAL: NCT02511457
Title: Validation of Measurement of Cardiac Output With LiDCO Rapid and TEE (Trans Esophageal Echocardiography) by Comparing With Intermittent Thermodilution Technique in Cardiac Surgical Patients
Brief Title: Comparison of Cardiac Output With LiDCO Rapid and TEE Against Thermodilution Technique in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Sudhakar Subramani, M.D., University of Iowa
Other Study IDs: 201205760
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Low Cardiac Output
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Measurement of the cardiac output is one of the important hemodynamic monitoring tools in cardiac surgery. It helps determine the type of medications needed to maintain optimal hemodynamic status in the entire perioperative period. Thermodilution method using pulmonary artery catheter is considered has the gold standard for the measurement of cardiac output. Investigators would like to compare the most popular minimally-invasive devices used to measure cardiac output using arterial waveform: LiDCO Rapid and TEE with the thermodilution method at various phases of the cardiac surgery.

DETAILED DESCRIPTION:
Measurement of the cardiac output is one of the important hemodynamic monitoring tools in cardiac surgery. It helps determine the type of medications needed to maintain optimal hemodynamic status in the entire perioperative period. Thermodilution method using pulmonary artery catheter is considered has the gold standard for the measurement of cardiac output, however over the past 10 to 15 years it has been questioned about its safety and efficacy. There has been a surge in recent years of less invasive devices capable of measuring cardiac output by various means, including bioimpedance, transpulmonary thermodilution, transthoracic and transesophageal echocardiography, and arterial waveform analysis.

There is a variety of devices currently available for cardiac output measurement by arterial-waveform analysis. These devices have been compared to each other, and to the pulmonary artery catheter as the gold standard. However, the companies manufacturing these devices have made software upgrades that they believe improves their performance. No studies have been performed comparing the uncalibrated arterial waveform based cardiac output measurement device,LiDCORapid since the software upgrades. In addition to baseline cardiac output measurements, Investigators intend to study the effect of volume loading (by trendelenburg position), sympathetic stimulus (incision), a vasodilated state (15 minutes after separation from CPB) and chest closure on cardiac output measured by the three different techniques.

In addition to cardiac output the investigators would like to measure stroke volume ,Systemic Vascular Resistance, stroke volume variation with LiDCO . The main purpose is to validate the accuracy of measurements by these two minimally-invasive methods in comparison with thermodilution method in various hemodynamic states.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac procedures other than those specified in the exclusion criteria

Exclusion Criteria:

* All emergency cardiac procedures, prisoners and pregnant women, patients who are scheduled for ventricular assist devices and those with severe aortic, mitral and tricuspid insufficiency will be excluded.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All elective adult cardiac surgery patients who are scheduled in UIHC from Sep 2012 to August 2015 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is measured cardiac output by LiDCO Rapid is as equivalent ( within 30%) as measured by pulmonary artery catheter using intermittent thermodilution method among patients undergoing elective cardiac surgery. | During intraoperative period.

SECONDARY OUTCOMES:
The secondary objective of the study is measured cardiac output by TEE using VTI at LVOT is as equivalent ( within 30%) as measured by pulmonary artery catheter using intermittent thermodilution method among patients undergoing elective cardiac surgery. | During intraoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Subramani, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Result] Hadian M, Kim HK, Severyn DA, Pinsky MR. Cross-comparison of cardiac output trending accuracy of LiDCO, PiCCO, FloTrac and pulmonary artery catheters. Crit Care. 2010;14(6):R212. doi: 10.1186/cc9335. Epub 2010 Nov 23. PMID 21092290
- [Result] Cecconi M, Dawson D, Casaretti R, Grounds RM, Rhodes A. A prospective study of the accuracy and precision of continuous cardiac output monitoring devices as compared to intermittent thermodilution. Minerva Anestesiol. 2010 Dec;76(12):1010-7. Epub 2010 Jul 16. PMID 20634793